CLINICAL TRIAL: NCT06255080
Title: Re-defining Proficiency Levels Might be Necessary When Virtual Reality Simulator Software is Updated - a Randomized Trial
Brief Title: Comparing Skills Acquisition on Different Laparoscopy Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Anishan Vamadevan, Research Fellow, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Software changes on LAPSIM
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Simulation Training; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group practiced the proficiency-based program on the LAPSIM(R) simulator using the new 2019-version of the software
  Interventions: Other: Training intervention
- Control Group (No Intervention): This group practiced the proficiency-based program on the LAPSIM(R) simulator using the original (and evidence based) 2016-version of the software

INTERVENTIONS:
Other: Training intervention — The intervention consists of making the intervention group practice till proficiency using the 2019-version.
  The control group practices till they have reached proficiency using the standard 2016-version.
  We wanted to compare time to completetion for the intervention. For the follow-up test we invited all participants to return after 4-6 weeks (where no training was allowed) and made them practice till proficiency again using the standard 2016-version. Time to reach proficiency for the follow-up test was compared.
  Arms: Intervention group

SUMMARY:
Simulation based training is a standard part of surgical training. Over the years virtual reality simulator have been more and more integrated into the surgical curriculum for surgical novices.

Evidence shows that practicing using proficiency-based training programs significantly reduces the operation time and complication rates for during intial operations for young doctors.

The aim of this trial is to examine if skills obtained on a newer software version is transferable to the original software.

ELIGIBILITY:
Inclusion Criteria:

* Medical students without any prior laparoscopy experience in both a clinical or simulated setting

Exclusion Criteria:

* Prior experience with simulation based laparoscopy or clinical experience with laparoscopy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Time to reach proficiency (in minutes) | 1-2 months
  To examine if there was any difference in the time to reach proficiency for the two software versions

SECONDARY OUTCOMES:
Transferability of skills | 2-3 weeks
  We made all 20 participants return for a follow-up test, where they had to practice till they reached proficiency again using the standard 2016-version. Time to complete was compared

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No